CLINICAL TRIAL: NCT00868660
Title: A Phase I, Double Blind, Placebo-Controlled Study of ZP1848 Administered as Subcutaneous Bolus Injections in Healthy Subjects Followed by Multiple Doses in Patients With Crohn's Disease in Remission
Brief Title: Healthy Normal Single Ascending Dose and Crohn's Patient Multiple Ascending Dose
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zealand Pharma (Industry)
Responsible Party: Christian Thorkildsen, Project Director, Zealand Pharma A/S
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZP08-216; AA75468; NCT01429922 (obsolete NCT alias)
Record Dates: First submitted 2009-03-23; First posted 2009-03-25 (Estimated); Last update posted 2010-11-02 (Estimated); Status verified 2010-11

CONDITIONS: Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ZP1848 (Experimental): Healthy Subjects or Crohn's Disease patients
  Interventions: Drug: ZP1848
- Placebo (Placebo Comparator): Healthy subjects or Crohn's Disease patients
  Interventions: Drug: ZP1848

INTERVENTIONS:
Drug: ZP1848 — sc. bolus

SUMMARY:
Healthy Normal Single Ascending Dose and Crohn's patient Multiple Ascending Dose

DETAILED DESCRIPTION:
A Phase I, Double blind, Placebo-controlled, safety and tolerability study of ZP1848 administered as Ascending single Dose, SUBCUTANEOUS bolus injections in healthy SUBJECTS followed by a Multiple Dose cohort of patients with stable Crohn's disease in remission

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male and/or females, 18 to 50 years of age
* Body mass index (BMI)18-30. Chrons Inclusion
* Adult male and/or females, 18 to 60 years of age (inclusive).
* Body mass index (BMI) ≥ 18 and ≤ 30 (kg/m2).
* Crohn's Disease Activity Index (CDAI) score < 150.
* In a stable state of Crohn's disease as per the Investigator's opinion.
* Free of steroid treatment (therapy targeted for the GI tract only) within the 3 months prior to Day 1.

Exclusion Criteria:

* History or presence of dysplasia, cancer, chronic hepatitis, HIV, tuberculosis (TB), or histoplasmosis.
* Fistula within the 3 months prior to dosing. 3. Ostomy (having ostomy now or at any time in the past). 4. Any surgery for the treatment of inflammatory bowel disease (IBD) within the 3 months prior to Day 1. 5. Short Bowel Syndrome (SBS). 6. Any other condition, chronic disease, or prior therapy, which in the opinion of the Investigator/Investigator's designee would put the patient at undue risk or would make the patient unsuitable for the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2009-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
safety and tolerability | January2009-January2010

SECONDARY OUTCOMES:
Pharmacokinetics | Jan 2009 - Jan 2010

CONTACTS AND LOCATIONS:
Overall Officials: Christian Thorkildsen, Study Director — Zealand Pharma A/S
Locations (1):
- CRI Worldwide, Willingboro, New Jersey, United States